CLINICAL TRIAL: NCT01931202
Title: Mechanisms of Antidepressant Non-Response in Late-Life Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Bret Rutherford, Assistant Professor of Clinical Psychiatry, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6836
Record Dates: First submitted 2013-08-26; First posted 2013-08-29 (Estimated); Results first posted 2020-04-08 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Double Blind-Placebo (Placebo Comparator): Blinded treatment with placebo, one pill a day. If after the 4 weeks, the patient has not remitted, they will be increased to 2 pills a day.
  Interventions: Drug: Placebo oral tablet
- Double Blind-Escitalopram (Active Comparator): Blinded treatment with either escitalopram 10mg, increased to escitalopram 20mg at week 4 if depression has not remitted.
  Interventions: Drug: Escitalopram
- Open Treatment with Escitalopram (Active Comparator): Open treatment with 10mg of escitalopram, increased to 20mg if depression has not remitted at week 4.
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — Escitalopram is an antidepressant of the selective serotonin reuptake inhibitor (SSRI) class. It is FDA approved for the treatment of major depressive disorder (MDD) and generalized anxiety disorder (GAD) in adults and children over 12 years of age.
  Other Names: Lexapro
  Arms: Double Blind-Escitalopram; Open Treatment with Escitalopram
Drug: Placebo oral tablet — Inert substance or treatment which is designed to have no therapeutic value but resemble the active medication in this study
  Other Names: placebo
  Arms: Double Blind-Placebo

SUMMARY:
This project seeks to elucidate the mechanisms by which antidepressant medications have limited efficacy in Late Life Depression (LLD) in order to develop new treatment interventions for this prevalent and disabling illness. Investigators hypothesize that the presence of executive dysfunction (ED),which is common in depressed adults over 60, impairs the ability to form appropriate expectancies of improvement with antidepressant treatment. Greater expectancy has been shown to improve antidepressant treatment outcome and is hypothesized to be a primary mechanism of placebo effects. Moreover, white matter hyperintensities (WMH) on magnetic resonance imaging (MRI) are more prevalent in patients with LLD compared to healthy controls. It has been argued that WMH contribute to the pathogenesis of LLD with ED and decrease the efficacy of antidepressant medications by disrupting connections between prefrontal cortical (PFC) and subcortical structures. Vascular lesions to white matter tracts may also compromise the pathway by which expectancy-based placebo effects influence depressive symptoms. Expectancies reflect activation in PFC areas that may improve depressive symptoms by modulating the activity of subcortical regions subserving negative affective systems (i.e., amygdala) as well as those important in reward and hedonic capacity (nucleus accumbens and ventral striatum). Thus, LLD patients with ED and WMH may sustain a "double-hit" to their ability to experience placebo effects in antidepressant treatments: ED diminishes the ability to generate appropriate treatment expectancies, while WMH disrupt the physiologic pathways by which expectancies lead to improvement in depressive symptoms.

DETAILED DESCRIPTION:
To determine whether decreased antidepressant medication response in LLD patients with ED and WMH is caused by a loss of expectancy effects, Investigators will evaluate 130 outpatients with LLD at baseline to determine their degree of ED (interference score on Stroop Color-Word Test), WMH burden (severity score on Fazekas modified Coffey Rating Scale derived from anatomical MRI), and white matter tract integrity (using diffusion tensor imaging [DTI]). Building on work from the investigators K23 Award, the investigator will manipulate participants' expectancy of improvement in an 8-week duration antidepressant trial by randomizing patients between open administration of escitalopram (i.e., high expectancy) and placebo-controlled administration of escitalopram (i.e., low expectancy). The difference in antidepressant response observed between open and placebo-controlled medication treatment is a measure of the expectancy contribution to outcome, which is substantial in younger depressed adults but investigators hypothesize this will be diminished in LLD patients with ED and WMH.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 60-90 years
* Diagnosis with nonpsychotic Diagnostic and Statistical Manual (DSM) IV MDD
* 24-item Hamilton Rating Scale for Depression (HRSD) score ≥ 16
* Willing to and capable of providing informed consent and complying with study procedures

Exclusion Criteria:

* Current comorbid Axis I DSM IV disorder other than Nicotine Dependence, Adjustment Disorder, or Anxiety Disorder
* diagnosis of substance abuse or dependence (excluding Nicotine Dependence) within the past 12 months
* History of psychosis, psychotic disorder, mania, or bipolar disorder
* Diagnosis of probable Alzheimer's Disease, Vascular Dementia, or Parkinson's Disease
* MMSE < 24
* HRSD suicide item > 2 or Clinical Global Impressions (CGI)-Severity score of 7 at baseline
* history of allergic or adverse reaction to escitalopram, or non-response to adequate trial of escitalopram (at least 4 weeks at dose of 20mg) during the current episode
* current treatment with psychotherapy, antidepressants, antipsychotics, or mood stabilizers
* having contraindication to MRI scanning (such as metal in body) or unable to tolerate the scanning procedures (i.e., severe obesity, claustrophobia)
* acute, severe, or unstable medical or neurological illness

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2014-02-19 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2020-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bret Rutherford, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wengler K, Ashinoff BK, Pueraro E, Cassidy CM, Horga G, Rutherford BR. Association between neuromelanin-sensitive MRI signal and psychomotor slowing in late-life depression. Neuropsychopharmacology. 2021 Jun;46(7):1233-1239. doi: 10.1038/s41386-020-00860-z. Epub 2020 Sep 12. PMID 32919398
- See also: Rutherford BR, Roose SP. A Model of Placebo Response in Antidepressant Clinical Trials. Am J Psychiatry. 2013 Jan 15. doi: 10.1176/appi.ajp.2012.12040474. [Epub ahead of print] PubMed PMID: 23318413 — https://www.ncbi.nlm.nih.gov/m/pubmed/23318413/?i=6&from=/17998306/related

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 138 subjects signed consent, 108 were randomized to one of the 3 arms therefore they cannot be classified to any of the below arms.
Groups:
- Double Blind-Placebo Group: Blinded treatment with placebo, one pill a day. If after the 4 weeks, the patient has not remitted, they will be increased to 2 pills a day.
- Double Blind-Escitalopram Group: Blinded treatment with escitalopram 10mg increased to escitalopram 20mg or placebo at week 4 if depression has not remitted
  Escitalopram: Escitalopram is an antidepressant of the selective serotonin reuptake inhibitor (SSRI) class. It is FDA approved for the treatment of major depressive disorder (MDD) and generalized anxiety disorder (GAD) in adults and children over 12 years of age.
Period: Overall Study
Arm/Group | Double Blind-Placebo Group | Double Blind-Escitalopram Group | Open Treatment With Escitalopram
Started | 8 | 51 | 49
Completed | 8 | 46 | 45
Not Completed | 0 | 5 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 5 | 2

BASELINE CHARACTERISTICS:
Population: Although 138 subjects were enrolled (signed consent), only 108 were randomized and included in analysis.
Groups:
- Placebo: Blinded treatment with placebo.
  Placebo oral tablet: Inert substance or treatment which is designed to have no therapeutic value but resemble the active medication in this study
- Escitalopram: Blinded treatment with either escitalopram, increased to escitalopram 20mg or placebo at week 4 if depression has not remitted
  Escitalopram: Escitalopram is an antidepressant of the selective serotonin reuptake inhibitor (SSRI) class. It is FDA approved for the treatment of major depressive disorder (MDD) and generalized anxiety disorder (GAD) in adults and children over 12 years of age.
- Total: Total of all reporting groups
Arm/Group | Placebo | Escitalopram | Open Treatment With Escitalopram | Total
Number analyzed (Participants) | 8 | 51 | 49 | 108
Age, Customized [Mean (Standard Deviation); unit: years]
  Age at Screening | 73.9 (7.2) | 70.7 (8.4) | 69.2 (7.2) | 70.2 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 32 | 32 | 70
  Male | 2 | 19 | 17 | 38
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 0 | 1 | 1
  Black/African American | 1 | 6 | 8 | 15
  White | 5 | 35 | 34 | 74
  More than one | 1 | 6 | 3 | 10
  Don't Know | 1 | 3 | 3 | 7
  Missing | 0 | 1 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 51 | 49 | 108
Hamilton Rating Scale for Depression (HRSD) [Mean (Standard Deviation); unit: units on a scale] — Our target is depressive symptomatology as measured by the Hamilton Rating Scale for Depression (HRSD). The HRSD is a 24-item questionnaire used as an indication of depression and a guide to evaluate recovery. Total scores range from 0-74, not including atypical symptoms sub-scale. A score of 16 or above is typically considered to indicate the presence of depressive symptoms. Higher scores indicate greater severity.
  units on a scale | 22.8 (4.9) | 23.6 (6.1) | 22.9 (6.3) | 23.2 (6.1)

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Rating Scale for Depression (HRSD)
Description: Our target is depressive symptomatology as measured by the Hamilton Rating Scale for Depression (HRSD). The HRSD is a 24-item questionnaire used as an indication of depression and a guide to evaluate recovery. Total scores range from 0-74, not including atypical symptoms sub-scale. A score of 16 or above is typically considered to indicate the presence of depressive symptoms. Higher scores indicate greater severity.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Double Blind-Escitalopram Group: Blinded treatment with escitalopram 10mg, increased to escitalopram 20mg at week 4 if depression has not remitted
  Escitalopram: Escitalopram is an antidepressant of the selective serotonin reuptake inhibitor (SSRI) class. It is FDA approved for the treatment of major depressive disorder (MDD) and generalized anxiety disorder (GAD) in adults and children over 12 years of age.
Arm/Group | Double Blind-Placebo Group | Double Blind-Escitalopram Group | Open Treatment With Escitalopram
Number analyzed (Participants) | 8 | 51 | 49
units on a scale | 22.8 (4.9) | 23.6 (6.1) | 22.9 (6.3)

2. Secondary Outcome: Hamilton Rating Scale for Depression (HRSD)
Description: as for outcome 1
Time Frame: Week 8
Population: Although 138 subjects were enrolled (signed consent) and 108 were randomized, only 99 completed the Hamilton Rating Scale for Depression (HRSD) at week 8.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Double Blind-Escitalopram Group: Blinded treatment with escitalopram 10mg , increased to escitalopram 20mg at week 4 if depression has not remitted
  Escitalopram: Escitalopram is an antidepressant of the selective serotonin reuptake inhibitor (SSRI) class. It is FDA approved for the treatment of major depressive disorder (MDD) and generalized anxiety disorder (GAD) in adults and children over 12 years of age.
Arm/Group | Double Blind-Placebo Group | Double Blind-Escitalopram Group | Open Treatment With Escitalopram
Number analyzed (Participants) | 8 | 46 | 45
units on a scale | 13.25 (5.50) | 14.39 (8.13) | 11.67 (7.58)

3. Secondary Outcome: Quick Inventory of Depressive Symptoms (QIDS-SR)
Description: QIDS-SR is a 16 item scale self-report form that was used to measure depression outcomes. This self-report is valuable in this study, because it is less susceptible to clinician and rater bias. The QIDS-SR has been increasingly used in antidepressant studies due to its equivalent weightings for each symptom item, clearly understandable anchor points, and inclusion of all DSM criteria for depression. The scores range from 0-27 with 27 being worse depressive symptoms.
Time Frame: Baseline
Population: 138 subjects were consented, of which 108 were randomized, however only 107 completed baseline Quick Inventory of Depressive Symptoms (QIDS-SR).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double Blind-Placebo Group | Double Blind-Escitalopram Group | Open Treatment With Escitalopram
Number analyzed (Participants) | 8 | 50 | 49
units on a scale | 12.4 (4.4) | 13.5 (4.5) | 13.0 (4.7)

4. Secondary Outcome: Quick Inventory of Depressive Symptoms (QIDS-SR)
Description: as for outcome 3
Time Frame: Week 8
Population: 138 subjects were consented, of which 108 were randomized, however only 99 completed week 8 Quick Inventory of Depressive Symptoms (QIDS-SR).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double Blind-Placebo Group | Double Blind-Escitalopram Group | Open Treatment With Escitalopram
Number analyzed (Participants) | 8 | 46 | 44
units on a scale | 8.00 (2.93) | 6.93 (5.14) | 6.34 (5.31)

5. Secondary Outcome: Credibility and Expectancy Scale-Better (CES)
Description: CES is an 8 item scale in which subjects rate their impression of the credibility of the treatment and how they estimate their expectation of improvement. The CES is the most widely used measure of expectancy and has demonstrated good psychometric properties in multiple studies. Question 2 ('Better') asks the patient the chances of their depression being completely better at the end of this study, from 1 = very poor to 7 = very good. The higher the number, the higher the expectancy that they will be better.
Time Frame: Pre-Baseline
Population: 138 subjects were consented, of which 108 were randomized, however only 101 completed pre-baseline Credibility and Expectancy Scale-Better (CES).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double Blind-Placebo Group | Double Blind-Escitalopram Group | Open Treatment With Escitalopram
Number analyzed (Participants) | 8 | 46 | 47
units on a scale | 6 (1.1) | 5.5 (1.2) | 5.3 (1.3)

6. Secondary Outcome: Credibility and Expectancy Scale-Better (CES)
Description: as for outcome 5
Time Frame: Week 0
Population: 138 subjects were consented, of which 108 were randomized, however only 106 completed week 0 Credibility and Expectancy Scale-Better (CES).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Double Blind-Escitalopram Group: Blinded treatment with either escitalopram 10mg , increased to escitalopram 20mg at week 4 if depression has not remitted
  Escitalopram: Escitalopram is an antidepressant of the selective serotonin reuptake inhibitor (SSRI) class. It is FDA approved for the treatment of major depressive disorder (MDD) and generalized anxiety disorder (GAD) in adults and children over 12 years of age.
Arm/Group | Double Blind-Placebo Group | Double Blind-Escitalopram Group | Open Treatment With Escitalopram
Number analyzed (Participants) | 8 | 50 | 48
units on a scale | 5.63 (0.92) | 5.00 (1.36) | 5.67 (1.40)

7. Secondary Outcome: Credibility and Expectancy Scale-Depression
Description: CES is an 8 item scale in which subjects rate their impression of the credibility of the treatment and how they estimate their expectation of improvement. The CES is the most widely used measure of expectancy and has demonstrated good psychometric properties in multiple studies. CES question 3 ('Depression') asks how the patient's depression will be at the end of the study, compared with now, from 1 = much worse to 7= much better. The higher the number, the higher the expectancy that their depression will be much better.
Time Frame: Pre-baseline
Population: 138 subjects were consented, of which 108 were randomized, however only 101 completed pre-baseline Credibility and Expectancy Scale-Depression.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double Blind-Placebo Group | Double Blind-Escitalopram Group | Open Treatment With Escitalopram
Number analyzed (Participants) | 8 | 46 | 47
units on a scale | 6.3 (1.2) | 6.0 (0.9) | 5.9 (0.9)

8. Secondary Outcome: Credibility and Expectancy Scale-Depression
Description: as for outcome 7
Time Frame: Week 0
Population: 138 subjects were consented, of which 108 were randomized, however only 106 completed week 0 Credibility and Expectancy Scale-Depression.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double Blind-Placebo Group | Double Blind-Escitalopram Group | Open Treatment With Escitalopram
Number analyzed (Participants) | 8 | 50 | 48
units on a scale | 5.88 (0.99) | 5.40 (1.09) | 6.06 (0.84)

9. Secondary Outcome: Quick Inventory of Depression Scale (QIDS-SR): Expectancy
Description: This 16-items assessment is used to rate the 9 criterion symptom domains of a major depressive episode: 4 items are used to rate sleep disturbance (early, middle, and late insomnia plus hypersomnia); 2 items are used to rate psychomotor disturbance (agitation and retardation); 4 items are used to rate appetite/weight disturbance (appetite increase or decrease and weight increase or decrease). Only 1 item is used to rate the remaining 6 domains (depressed mood, decreased interest, decreased energy, worthlessness/guilt, concentration/decision making, and suicidal ideation). Each item is rated 0-3. For symptom domains that require more than 1 item, the highest score of the item relevant for each domain is taken. The total score ranges from 0-27. A lower rating indicates higher expectancy of improvement and lower expectation of depressive symptomatology, and a higher rating indicates lower expectancy of improvement, higher expectation of depression.
Time Frame: Pre-Baseline
Population: 138 subjects were consented, of which 108 were randomized, however only 101 completed pre-baseline Quick Inventory of Depression Scale (QIDS-SR): Expectancy.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double Blind-Placebo Group | Double Blind-Escitalopram Group | Open Treatment With Escitalopram
Number analyzed (Participants) | 8 | 46 | 47
units on a scale | 5.3 (6.2) | 4.8 (3.7) | 5.8 (4.5)

10. Secondary Outcome: Quick Inventory of Depression Scale (QIDS-SR): Expectancy
Description: as for outcome 9
Time Frame: Week 0
Population: 138 subjects were consented, of which 108 were randomized, however only 107 completed week 0 Quick Inventory of Depression Scale (QIDS-SR): Expectancy.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double Blind-Placebo Group | Double Blind-Escitalopram Group | Open Treatment With Escitalopram
Number analyzed (Participants) | 8 | 50 | 49
units on a scale | 6.63 (3.42) | 6.20 (4.83) | 4.92 (3.83)

11. Secondary Outcome: Executive Dysfunction: Stroop Color Word
Description: Stroop Color Word test asks patients to name the color of a word rather than reading the word. Stroop Color Word is how many colors they can name in 45 sec (higher is better, e.g., less executive dysfunction).
Time Frame: Pre-Baseline
Population: 138 subjects were consented, of which 108 were randomized, however only 106 completed pre-baseline Executive Dysfunction: Stroop Color Word.
Measure: Mean (Standard Deviation); unit: correct items
Arm/Group | Double Blind-Placebo Group | Double Blind-Escitalopram Group | Open Treatment With Escitalopram
Number analyzed (Participants) | 7 | 50 | 49
correct items | 31.7 (6.1) | 31.0 (9.0) | 32.6 (11.0)

12. Secondary Outcome: Executive Dysfunction: Stroop Interference
Description: The Stroop is a measure of inhibition under distracting conditions that is sensitive to frontal lobe dysfunction. in Stroop Color Word test patients are to name the color of a word rather than reading the word. Stroop Color Word is how many colors they can name in 45 sec (higher is better, e.g., less executive dysfunction). Stroop Interference is this score adjusted for age and education.
Time Frame: Pre-Baseline
Population: 138 subjects were consented, of which 108 were randomized, however only 105 completed pre-baseline Executive Dysfunction: Stroop Interference.
Measure: Mean (Standard Deviation); unit: correct items
Arm/Group | Double Blind-Placebo Group | Double Blind-Escitalopram Group | Open Treatment With Escitalopram
Number analyzed (Participants) | 6 | 50 | 49
correct items | 42.2 (6.8) | 42.9 (11.2) | 44.1 (10.4)

13. Secondary Outcome: White Matter Hyperintensity (WMH) Outcome- Total WMH
Description: Magnetic Resonance Imaging (MRI) of the Brain was acquired. We rated the severity of WMH on axial T2 FLAIR images using the Fazekas modified Coffey Rating Scale. Deep WMH are scored as 0 (absent), 1 (punctate foci), 2 (beginning confluence of foci), and 3 (large confluent areas); subcortical gray matter HIs (basal ganglia) are scored as 0 (absent), 1 (punctate), 2 (multipunctate), and 3 (diffuse); periventricular HIs are scored as 0 (absent), 1 (caps), 2 (smooth halo), and 3 (irregular and extending into the deep white matter). Our primary measure of WMH burden will be DWMH score, which has been used to establish the only empirically validated diagnostic criteria for vascular depression, where scores of 0-1 were normal, but 2-3 indicated WHM.
Time Frame: Pre-Baseline
Population: 138 subjects signed consent and 108 were randomized, however not all participants underwent MRI scanning.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Double Blind-Escitalopram Group: Blinded treatment with either escitalopram 10mg o increased to escitalopram 20mg at week 4 if depression has not remitted
  Escitalopram: Escitalopram is an antidepressant of the selective serotonin reuptake inhibitor (SSRI) class. It is FDA approved for the treatment of major depressive disorder (MDD) and generalized anxiety disorder (GAD) in adults and children over 12 years of age.
Arm/Group | Double Blind-Placebo Group | Double Blind-Escitalopram Group | Open Treatment With Escitalopram
Number analyzed (Participants) | 5 | 28 | 33
score on a scale | 2.3 (1.7) | 2.1 (1.9) | 1.9 (2.2)

ADVERSE EVENTS:
Time Frame: Adverse events were collected through the 8 week period of the study.
Description: Adverse events were collected during weekly visit with the patients.
Groups:
- Double Blind-Placebo Group: Blinded treatment with placebo, 1 pill a day for 4 weeks. At week 4, if patients have not remitted, they were increased to 2 pills a day.
- Double Blind-Escitalopram Group: Blinded treatment with either escitalopram 10mg, increased to escitalopram 20mg at week 4 if depression has not remitted
  Escitalopram: Escitalopram is an antidepressant of the selective serotonin reuptake inhibitor (SSRI) class. It is FDA approved for the treatment of major depressive disorder (MDD) and generalized anxiety disorder (GAD) in adults and children over 12 years of age.
Arm/Group | Double Blind-Placebo Group | Double Blind-Escitalopram Group | Open Treatment With Escitalopram
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/51 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/8 | 2/51 | 1/49
Other Adverse Events (participants affected / at risk) | 0/8 | 0/51 | 0/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double Blind-Placebo Group (N=8) | Double Blind-Escitalopram Group (N=51) | Open Treatment With Escitalopram (N=49)
Fall (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Chest Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-08-22): https://cdn.clinicaltrials.gov/large-docs/02/NCT01931202/Prot_000.pdf
  • Statistical Analysis Plan (2013-02-05): https://cdn.clinicaltrials.gov/large-docs/02/NCT01931202/SAP_001.pdf